CLINICAL TRIAL: NCT01724450
Title: Carvedilol Effect in Preventing Chemotherapy - Induced Cardiotoxicity. A Randomized Double Blind Study.
Brief Title: Carvedilol Effect in Preventing Chemotherapy - Induced Cardiotoxicity
Acronym: Ceccy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Hospital A.C. Camargo (Other); Instituto do Cancer do Estado de São Paulo (Other)
Responsible Party: Principal Investigator, Edimar Alcides Bocchi, phd, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Ceccy Trial
Record Dates: First submitted 2012-06-11; First posted 2012-11-09 (Estimated); Last update posted 2018-02-05 (Actual); Status verified 2018-01

CONDITIONS: Breast Cancer; Heart Failure; Cardiotoxicity
Keywords: Breast Cancer; Heart Failure; Cardiotoxicity; Biomarkers
MeSH Terms: conditions — Breast Neoplasms; Heart Failure; Cardiotoxicity | interventions — Carvedilol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Carvedilol (Active Comparator)
  Interventions: Drug: Carvedilol
- Control (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Carvedilol — 50mg/day for 24 weeks. The dose of carvedilol will be up titrate before the dose of 50mg/day
  Arms: Carvedilol
Drug: Placebo — Placebo similar to the carvedilol up titration but wit no active drug.
  Arms: Control

SUMMARY:
The purpose of this study is to evaluate if carvedilol can prevent the cardiotoxicity after chemotherapy in breast cancer.

DETAILED DESCRIPTION:
Dilated cardiomyopathy secondary to chemotherapy accounts for approximately 1% of all dilated cardiomyopathies.

Initial studies showed beneficial effect of the use of carvedilol for the prevention of chemotherapy-induced cardiomyopathy. This study has the objective to evaluate the effectiveness of carvedilol for the prevention of chemotherapy-induced cardiomyopathy. Will be selected 200 patients referred for chemotherapy that includes anthracyclines for breast cancer.These patients will be randomized to carvedilol or placebo and will have periodic assessment of cardiac function with echocardiography and biomarkers until complete chemotherapy and 24 months later.

ELIGIBILITY:
Inclusion Criteria:

Patients diagnosed with breast cancer, with an indication of chemotherapy that includes anthracycline.

Exclusion Criteria:

Failure analysis of ventricular function; History of chemotherapy or radiotherapy; Previous symptoms of heart failure; Presence of cardiomyopathy; Presence of Coronary Artery Disease; Aortic valve disease or moderate to severe mitral regurgitation; Contraindication to the use of β-blocker; Use of inhibitors of angiotensin converting enzyme, angiotensin receptor blockers or β-blockers.

Patients with HER 2 expression

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Prevention of systolic dysfunction in patients undergoing chemotherapy with anthracycline. Systolic dysfunction is characterized by a 10% drop in ejection fraction of left ventricle. | 96 weeks

SECONDARY OUTCOMES:
Prevention of myocardial injury measured by the levels of biomarkers (ultrasensitive troponin, BNP and miRNA-208) Effect of carvedilol in the prevention of diastolic dysfunction. | 96 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Edimar Alcides Bocchi, PHD, Principal Investigator — Heart Institute of University of Sao Paulo
Locations (1):
- Heart Institute University of Sao Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Wanderley MRB Jr, Avila MS, Fernandes-Silva MM, Cruz FDD, Brandao SMG, Rigaud VOC, Hajjar LA, Filho RK, Cunha-Neto E, Bocchi EA, Ayub-Ferreira SM. Plasma biomarkers reflecting high oxidative stress in the prediction of myocardial injury due to anthracycline chemotherapy and the effect of carvedilol: insights from the CECCY Trial. Oncotarget. 2022 Jan 25;13:214-223. doi: 10.18632/oncotarget.28182. eCollection 2022. PMID 35087624
- [Derived] Avila MS, Ayub-Ferreira SM, de Barros Wanderley MR Jr, das Dores Cruz F, Goncalves Brandao SM, Rigaud VOC, Higuchi-Dos-Santos MH, Hajjar LA, Kalil Filho R, Hoff PM, Sahade M, Ferrari MSM, de Paula Costa RL, Mano MS, Bittencourt Viana Cruz CB, Abduch MC, Lofrano Alves MS, Guimaraes GV, Issa VS, Bittencourt MS, Bocchi EA. Carvedilol for Prevention of Chemotherapy-Related Cardiotoxicity: The CECCY Trial. J Am Coll Cardiol. 2018 May 22;71(20):2281-2290. doi: 10.1016/j.jacc.2018.02.049. Epub 2018 Mar 11. PMID 29540327